CLINICAL TRIAL: NCT02210026
Title: A Study to Evaluate the Efficacy of Seattle-PAP for the Respiratory Support of Premature Infants
Brief Title: Seattle-PAP Bubble Nasal CPAP and Work of Breathing
Acronym: Seattle-PAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Charles Smith, Professor, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Seattle-PAP 001
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Respiratory Distress Syndrome In Premature Infants; Bronchopulmonary Dysplasia; Newborn Primary Sleep Apnea
Keywords: bubble nasal continuous positive airway pressure (Bn-CPAP); work of breathing; pressure-rate products
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Bronchopulmonary Dysplasia; Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Infants will be assessed on standard bubble nasal CPAP, then on Seattle-PAP bubble nasal CPAP, then again on standard bubble nasal CPAP.
  Interventions: Device: Seattle-PAP

INTERVENTIONS:
Device: Seattle-PAP — We propose to test the hypothesis that by introduction of variation in airway pressure Seattle bubble nasal continuous positive airway pressure (Seattle-PAP) reduces work of breathing in very low birth weight infants more effectively than standard bubble nasal continuous positive airway pressure.
  Other Names: Sea-PAP

SUMMARY:
The investigators propose to test the hypothesis that Seattle bubble nasal continuous positive airway pressure (Seattle-PAP) supports respiratory physiology in very low birth weight (VLBW) infants more effectively than standard bubble nasal continuous positive airway pressure.

DETAILED DESCRIPTION:
The primary outcome variable is work of breathing (WOB) over a two hour period, estimated from pressure-rate products, which are assessed with 6 Fr (2 mm) catheters placed in the distal esophagus for monitoring esophageal pressures (Pes), thereby estimating changes in pleural pressures during breath cycles. The following endpoints would also be assessed: Oxygen saturations and Fraction of Inspired Oxygen (FiO2) needed to keep saturations in acceptable ranges, Heart Rates (HR), transcutaneous carbon dioxide (TcPCO2), and respiratory rates throughout the 6 hour study period.

Objective determination of when an infant requires more or less respiratory support is difficult, but measurements of pressure-rate products as estimates of work of breathing, using esophageal catheters, can estimate an infant's respiratory effort. However, objective, simple-to-use, low cost, and non-invasive methods and tools to determine an infant's respiratory effort do not exist currently.

This study also is designed to test the hypothesis that infants' chest and abdominal movements can be assessed quantitatively from video images in ways that can be correlated with intrathoracic pressures, as measured with esophageal catheters.

ELIGIBILITY:
Inclusion Criteria:

* infant born less than 32 weeks gestation
* admitted to texas pavilion for women
* between 6 and 72 hours post delivery
* stable on standard bubble nasal CPAP
* informed consent

Exclusion Criteria:

* major congenital anomalies or suspected chromosomal anomalies

Ages: 6 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Work of Breathing | Six hours
  The primary outcome variable is work of breathing (WOB) over three two hour periods, estimated from pressure-rate products, which are assessed with 6 Fr (2 mm) catheters placed in the distal esophagus for monitoring esophageal pressures (Pes), thereby estimating changes in pleural pressures during breath cycles.

SECONDARY OUTCOMES:
Video Recordings of Chest and Abdomen Movements during Breathing | Six hours
  This study also is designed to test the hypothesis that infants' chest and abdominal movements can be assessed quantitatively from video images in ways that can be correlated with intrathoracic pressures, as measured with esophageal catheters.

OTHER OUTCOMES:
FiO2 | Six hours
  Fraction of Inspired Oxygen (FiO2) needed to keep oxygen saturations in acceptable ranges will be assessed throughout the 6 hour study period.
Heart Rates | Six hours
  Heart rates will be assessed during the study period.
Transcutaneous Carbon Dioxide Levels | Six hours
  Transcutaneous carbon dioxide (TcPCO2) levels will be assessed.
Respiratory Rates | Six hours
  Respiratory rates will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Charles V Smith, PhD, Study Director — Seattle Children's Hospital; Stephen E Welty, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States